CLINICAL TRIAL: NCT02467803
Title: Shoulder Functional Outcomes of Patients With Proximal Humerus Fractures: Comparison of Two Different Treatment Protocol
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, HANDE GUNEY, PhD, Hacettepe University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: GO13/55
Record Dates: First submitted 2015-05-26; First posted 2015-06-10 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-05

CONDITIONS: Humeral Fracture
Keywords: humeral fracture; exercise; musculoskeletal manipulations
MeSH Terms: conditions — Humeral Fractures; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Intervention (Active Comparator): We applied scapula mobilization with shoulder ROM exercises
  Interventions: Other: Scapula mobilization; Other: Shoulder ROM exercises
- Control (Other): We applied only shoulder ROM exercises
  Interventions: Other: Shoulder ROM exercises

INTERVENTIONS:
Other: Scapula mobilization
  Arms: Intervention
Other: Shoulder ROM exercises

SUMMARY:
Fractures of the proximal humerus and the humeral head are most common injuries and the management is challenging. Functional therapy with short immobilization, followed by an accelerated physiotherapy protocol, is a simple, convenient, noninvasive, and efficient management option. This prospective randomized study is aim to assess the function of the upper extremity of patients who will be assigned to nonoperative treatment of a proximal humeral fracture. The primary objective is the Constant score. Secondary objectives are the Disabilities of the Arm, Shoulder, and Hand (DASH) instrument, measurement of shoulder range of motion (ROM), pain and depression level with Beck Depression Scale.

DETAILED DESCRIPTION:
In this prospective randomized controlled trial, informed consent forms were obtained from all participants and they were informed about the study based on the Declaration of Helsinki. The study was approved by local ethics committee of Hacettepe University (GO13/55). After comprehensive clinical evaluation, subjects were randomly assigned to the intervention group or the control group, using Random Allocation Software. The intervention group received scapular mobilization with upper extremity ROM exercises, the control group received only shoulder ROM exercises.

Patients with a radiographically proven, closed fracture of the proximal humerus admitted to the emergency department of Hacettepe University Hospital, who were considered suitable for primary nonoperative management by the orthopedic surgeon on charge, were asked to participate in this investigation.

The exclusion criteria are (1) skeletally immature patients (2) patients presenting to the hospital 10 days or more after injury (3) patients with open fractures or multiple trauma (4) pre-existing illness affecting the function of the upper limb, such as multiple sclerosis, paraplegia, and others (5) patients with a history of drug or alcohol abuse (6) patients with cooperation problems or problems in attending all scheduled study visits.

Patients' demographics (ie, gender, age, profession, smoking, concomitant diseases, medication) and injury characteristics (ie, accident type, energy level of trauma, concomitant injuries, fracture classification) will be recorded. Patients will be asked to rate their upper limb function 1 week before the accident to determine their baseline DASH score using the extended 3-modular questionnaire.13 Normalized DASH scores range from 0 (perfect function) to 100 (functionless extremity/joint).

Radiographs will be obtained in anterior-posterior projection and Neer's view upon admission in the emergency department and after manipulation. Additional computed tomography (CT) scans will be ordered at the discretion of the treating surgeon. Fractures were classified according to the American Orthopedics and Neer scheme by the orthopedic surgeon.

The intervention group will receive scapular mobilization after the sling will be removed. Scapular mobilization will be applied 3 times a week, a total of 24 sessions for 8 weeks. Each session lasted around 15-20 minutes. The shoulder flexion and abduction ROM exercises will be showed to the patients and performed 3 times, 10 sets on each day after the sling will be removed.

The control group will only perform the shoulder ROM exercises. Patients will be monitored and physically examined on the day sling removed (approximately 4 week after injury), 3 and 6 months after injury. Primary outcome measures comprised raw Constant scores and differences to the contralateral, healthy shoulder. The Constant score will show the change from baseline in shoulder functional outcomes at 6 months after injury) Pain levels will be measured on a 0-10 cm (0=no pain, 10=severe pain) visual analogue scale (VAS). The Constant score, DASH, pain level, shoulder ROM and Beck Depression Scale will be recorded on the day sling removed and 6 months after injury. Plain radiographs of the injured shoulder in 2 planes were obtained to determine fracture healing.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be recruited if they have radiologically proven, closed fracture of the humerus according to American Orthopedics and Neer classification.

Exclusion Criteria:

* skeletally immature patients
* patients presenting to the hospital 10 days or more after injury
* patients with open fractures or multiple trauma
* pre-existing illness affecting the function of the upper limb, such as multiple sclerosis, paraplegia, and others
* patients with a history of drug or alcohol abuse
* patients with cooperation problems or problems in attending all scheduled study visits.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Constant Score | Patients will be followed for 6 months. The differences between baseline score and at the end of 6 months score will be assessed.

REFERENCES:
- [Derived] Handoll HH, Elliott J, Thillemann TM, Aluko P, Brorson S. Interventions for treating proximal humeral fractures in adults. Cochrane Database Syst Rev. 2022 Jun 21;6(6):CD000434. doi: 10.1002/14651858.CD000434.pub5. PMID 35727196